CLINICAL TRIAL: NCT06904768
Title: A Cross-Over Study on the Effect of Shoulder Sling Use on Balance and Functional Mobility in Patients With Hemiplegia During the Subacute Phase of Stroke Rehabilitation
Brief Title: Effect of Shoulder Sling Use on Balance and Mobility in Subacute Stroke Patients
Acronym: SLS-Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arnaoutis Stylianos (Other)
Collaborators: University of West Attica (Other)
Responsible Party: Sponsor-Investigator, Arnaoutis Stylianos, Principal Investigator, University of West Attica
Organization: University of West Attica (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: SLS2025-GR01
Record Dates: First submitted 2025-03-23; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Hemiplegia; Balance Disorders; Mobility Limitation; Shoulder Subluxation; Stroke
Keywords: Stroke; Hemiplegia; mobility; dynamic balance; balance; shoulder brace; arm sling
MeSH Terms: conditions — Hemiplegia; Mobility Limitation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shoulder Sling (Experimental): Participants perform balance and mobility tests (TUG, FRT, mFSST) while wearing a shoulder sling on the affected upper limb.
  Interventions: Device: Shoulder Sling
- No Sling (Active Comparator): The same functional tests are performed without the use of a shoulder sling.
  Interventions: Other: No Sling

INTERVENTIONS:
Device: Shoulder Sling — Use of a shoulder sling (Reh4mat AM-SOB) on the affected upper limb during mobility and balance testing.
  Arms: Shoulder Sling
Other: No Sling — Functional mobility tests performed without the use of any assistive shoulder device.
  Arms: No Sling

SUMMARY:
This study examines whether wearing a shoulder sling can improve balance and mobility in people who are recovering from a stroke. Participants will perform simple movement and balance tests twice-once with the sling and once without. The goal is to find out if using the sling helps patients feel more stable and safe during walking and everyday activities.

DETAILED DESCRIPTION:
This is a cross-over study designed to evaluate the impact of shoulder sling use on balance and functional mobility in patients recovering from stroke in the subacute phase. Participants will be asked to complete three validated functional tests: the Timed Up and Go (TUG) test, the Functional Reach Test (FRT), and the Modified Four Square Step Test (mFSST). Each test will be performed twice, once with the shoulder sling and once without, in randomized order. The study aims to determine whether the sling provides measurable benefits in stability and performance during movement tasks. Data will be collected in rehabilitation centers under the supervision of clinical researchers.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke in the subacute phase (up to 6 months post-onset)
* Hemiplegia affecting one upper limb
* Brunnstrom stage < 4 for the affected upper limb
* Functional Ambulation Category (FAC) score > 3
* Age between 40 and 80 years
* Ability to follow simple instructions
* Medically stable to participate in balance and mobility testing
* Signed informed consent

Exclusion Criteria:

* Severe cognitive impairment (e.g. MMSE < 23)
* Visual or vestibular disorders affecting balance
* Significant orthopedic or musculoskeletal conditions of the lower limbs
* Uncontrolled cardiovascular or pulmonary disease
* Use of assistive devices that prevent sling application
* Severe aphasia interfering with understanding or communication
* Skin lesions or injuries at the shoulder region preventing sling use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) Test | Within 1 day (each participant performs it twice - with and without sling)
  Time required (in seconds) to stand up from a chair, walk 3 meters, turn, walk back, and sit down.
Functional Reach Test (FRT) | Within 1 day (each participant performs it twice - with and without sling)
  Distance reached (in centimeters) while standing and reaching forward without losing balance.
Modified Four Square Step Test (mFSST) | Within 1 day (each participant performs it twice - with and without sling)
  Time required to step in all four quadrants in a specified sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Chrysagis, Study Chair — University of West Attica
Locations (1):
- Filoktitis Recovery and Rehabilitation Center, Koropí, Attica, Greece

IPD SHARING:
Plan to Share IPD: No